CLINICAL TRIAL: NCT02641860
Title: A Phase I, Randomized, Single-centered, Double-blinded Clinical Trial of Allogenic Adipose Tissue-Derived Mesenchymal Progenitor Cells Therapy for Knee Osteoarthritis
Brief Title: Clinical Trial of Allogenic Adipose Tissue-Derived Mesenchymal Progenitor Cells Therapy for Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBMG-Allo-KOA-1.1
Record Dates: First submitted 2015-12-21; First posted 2015-12-30 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mesenchymal progenitor cells Dosage 1 (Other): Mesenchymal progenitor cells low-dose group
  Interventions: Biological: Mesenchymal progenitor cells
- Mesenchymal progenitor cells Dosage 2 (Other): Mesenchymal progenitor cells mid-dose group
  Interventions: Biological: Mesenchymal progenitor cells
- Mesenchymal progenitor cells Dosage 3 (Other): Mesenchymal progenitor cells high-dose group
  Interventions: Biological: Mesenchymal progenitor cells

INTERVENTIONS:
Biological: Mesenchymal progenitor cells — Biological: Allogenic Adipose tissue-derived mesenchymal progentior cells administrated for intra-articular use

SUMMARY:
Evaluate the safety and efficacy of Allogenic Adipose Tissue-Derived Mesenchymal Progenitor Cells Therapy for Knee Osteoarthritis.

DETAILED DESCRIPTION:
A Phase I, Randomized, Single-centered, Double-blinded Clinical Trial of Allogenic Adipose Tissue-Derived Mesenchymal Progenitor Cells Therapy for Knee Osteoarthritis.

This is a randomized,single-blind, double-blinded,phase I clinical trial. Subjects who are with a clinical diagnosis of knee osteoarthritis cartilage defects and will be randomly distributed 1:1:1 to different dosage group after signing the ICF and screening tests.The treatment will accept Allogenic ReJoinTM at the first and fourth week.The duration of the therapy is 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Object has an allergic history or is of an allergic constitution.
* Subjects who understand and sign the consent form for this study.
* Age: 18-70, males and females.
* Clinical diagnosis of degenerative arthritis by Radiographic Criteria of KellgrenLawrence:Duration of pain over Grade 4(11-point numeric scale)> 4 months.
* Course of Knee osteoarthritis:6 months to 10 years;
* The VAS score :3-8 points.(the data acquisition time is to stop using all analgesic at least 3 days ).

Exclusion Criteria:

* The subject has an allergic history of medicine or food。.
* The subject'BMI is over 30.
* The subject has uncontrolled or hard-to-control diseases of cardiovascular, liver, kidney or lung， endocrine system.
* The subject has an history malignant tumour.
* The subject has complications or diseases of: systemic or rheumatoid arthritis, Chondrocalcinosis articularis， Hemochromatosis，inflammatory arthropathy，avascular necrosis of femoral head，Paget's disease，hemophilic arthropathy，infectional arthritis，Charcot's disease，villonodular synovitis or synovial chondromatosis.
* The subject has severe generalized infectious diseases or local knee infection in the 3 months prior to this trial.
* The subject has disease of lower limbs which may be interfered knee evaluation, for example fibromyalgia, osphyalgia, lumbar disc protrusion and so on.
* The subject has coagulation disorders.
* The subject has received arthroscopic surgery or intra-articular operations in the 6 months prior to this trial.
* The subject has received other intra-articular injections for KOA in the 6 months preceding the trial.
* The subject has received aminoglucose or chondroitin sulfate in the 6 months preceding the trial.
* The subject has plan of knee prosthesis within the trial.
* The subject has contraindication of MRI, included but not only: the subject installed heart pacemaker、defibrillator、heart bracket、heart valve prosthesis、metal clip after aneurysm surgery、drug infusion device implanted in vivo、any electronic device implanted in the body（nerve stimulator、bone growth stimulator）、endovascular coil、strainer、ECG monitor、metal suture、shrapnel or sand of body, plate fixation and steel nail after fracture

  - Page 4 of 4 [DRAFT] - surgery、artificial limb or joint、audiphone、artificial cochlea、middle ear shift plant、metallic intraocular foreign body etc； claustrophobia、pregnancy within 3 months、critically ill patients.
* The subject tests positive for: HIV, hepatitis virus, syphilis or other infectious diseases.
* The subject has history of alcoholism, drug abuse, or mental illness in the 3 years prior to this trial.
* The subject has participated in any other clinical trial in the 3 months prior to this trial.
* The subject is pregnant, lactating or planning to conceive within the next 6 months.
* The subject has any other unsuitable or adverse condition to be determined by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety, recording of Adverse Events and Serious Adverse Events | 12 weeks,48 weeks
WOMAC Score | 48 weeks

SECONDARY OUTCOMES:
VAS Score | 48 weeks
SF-36 | 48 Weeks
The volume of articular cartilage | 48 weeks
WORMS Score | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology,Ren Ji Hospital,School of Medicine,Shanghai Jiao Tong University,Shanghai,China, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhao X, Ruan J, Tang H, Li J, Shi Y, Li M, Li S, Xu C, Lu Q, Dai C. Multi-compositional MRI evaluation of repair cartilage in knee osteoarthritis with treatment of allogeneic human adipose-derived mesenchymal progenitor cells. Stem Cell Res Ther. 2019 Oct 21;10(1):308. doi: 10.1186/s13287-019-1406-7. PMID 31639063